CLINICAL TRIAL: NCT06219304
Title: Evaluation of the Impact of Experimentally Induced Fatigability on Motor and Cognitive Functions. Effect of High Intensity Training on Motor and Cognitive Functions:a Pilot Randomized Controlled Trial
Brief Title: Effect of High Intensity Training on Motor and Cognitive Functions
Acronym: FAST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Ente Ospedaliero Ospedali Galliera (Other); Fondazione Italiana Sclerosi Multipla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FISM_FAST
Record Dates: First submitted 2023-09-22; First posted 2024-01-23 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Multiple Sclerosis
Keywords: fatigue; balance
MeSH Terms: conditions — Multiple Sclerosis; Fatigue

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multimodal functional training (Experimental): Multimodal training to reduce fatigue and to improve balance and strength
  Interventions: Other: Multimodal functional training
- Usual care (Active Comparator): Rehabilitative intervention to improve balance and mobility
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Multimodal functional training — 40 minutes of multimodal functional training: 20 minutes of aerobic training on treadmill, 10 minutes of dynamic balance training; 10 minutes of functional strength training.
  Arms: Multimodal functional training
Other: Usual care — Exercises aimed at improving balance and mobility
  Arms: Usual care

SUMMARY:
Fatigability is one of the most prevalent disorder in MS followed by walking, balance and cognitive disorders.

However, there are few experimental studies on the effects of fatigability on balance and gait hampering the knowledge of causal fatigue-related changes of walking, balance and cognition. Nowadays, instrumented systems such as wearable devices and optoelectronic systems are available and can be used to provide quantitative and objective indexes useful to monitor the changes of gait parameters during a fatiguing performance. (Moreover), instrumented assessment of patients' performances in dual task paradigms can reveal the possible impact of fatigability on cognitive functions. So far, high intensity functional training has been already used in MS to reduce fatigability. However, the true impact of reduced fatigability on walking, balance and cognition has not been assessed after a fatiguing task making impossible to understand the real impact of treatments focusing on fatigability on these functions.

Thus, the aims of the present proposal are to assess the: 1) the acute effect of experimentally induced motor fatigability on walking, balance and cognitive functions using an objective instrumented assessment before, during, and after an overground fatiguing walking test. 2) to investigate the effect of high intensity multimodal functional training to improve motor and cognitive disorders.

ELIGIBILITY:
Inclusion Criteria:

* More than 18 years of age
* Clinical diagnosis of Multiple Sclerosis (MS)
* Stable disease course without worsening more than 1 EDSS point over the last 3 months, -EDSS between 1.5 and 6 points
* Must be able to maintain upright posture without any assistance for 30 seconds
* Must be able to release a written informed consent.

Exclusion Criteria:

* MS relapse within the previous three months;
* Unable to comprehend the aims of the study and to follow test instructions;
* Diagnosis of major depression (DSM-5);
* Severe joint and/or bone disorders interfering with balance and gait (based upon clinical judgment);
* Cardiovascular diseases;
* Unconfirmed or uncertain diagnosis of MS (McDonald criteria)
* Other concomitant neurological disease;
* Patients already performing aerobic or walking exercise.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
difference in walking velocity during the fatiguing walking test | Baseline and at 6-8 weeks (after the completion of 16 training sessions)
  difference between velocity at the beginning of the test and velocity at the end of the fatiguability walking test, [m/s]

SECONDARY OUTCOMES:
gait asymmetry and gait regularity | Baseline and at 6-8 weeks (after the completion of 16 training sessions)
  gait asymmetry, gait regularity on the vertical and medio-lateral plane estimated by autocorrelation coefficients during the fatiguability walking test. These variables will be calculated from IMU's data.
Antero-posterior and medio-lateral accelerations in stabilometric tasks | Baseline and at 6-8 weeks (after the completion of 16 training sessions)
  Antero-posterior and medio-lateral accelerations from the IMU placed on the pelvis during a 60 seconds tasks performed with open and closed eyes.
Brief International Cognitive Assessment in Multiple Sclerosis (BICAMS) | Baseline and at 6-8 weeks (after the completion of 16 training sessions)
  BICAMS includes the Symbol Digit Modalities test (SDMT), the California Verbal Learning Test-2 (CVLT2) and the Brief Visuospatial Memory Test-Revised (BVMT-R).
  The total scores will be calculated considering the normative scores. The score on the oral SDMT varies from 0 to 110 and must be calculated with respect to years of schooling. The CVLT2 score varies from a minimum of 0 to a maximum of 16 points. The BVMT-R score ranges from a minimum of 0 to a maximum of 36 points.

OTHER OUTCOMES:
Modified Fatigue Impact Scale (MFIS) | Baseline and at 6-8 weeks (after the completion of 16 training sessions)
  Assessment of fatigue with a 21-items questionnaire that ranges from 0 to 36 as maximum score.
Multiple Sclerosis Walking Scale-12 (MSWS-12) | Baseline and at 6-8 weeks (after the completion of 16 training sessions)
  Assessment of perceived walking ability with a 12-items questionnaire that ranges from a minimum of 12 points to a maximum of 60 points.
Activities Balance Confidence Scale (ABC) | Baseline and at 6-8 weeks (after the completion of 16 training sessions)
  Assessment of perceived balance with a 16-items questinnaire that ranges from a minimum of 0% to a maximum of 100%.
Beck Depression Inventory (BDI-II). | Baseline and at 6-8 weeks (after the completion of 16 training sessions)
  Assessment of mood and anxiety with a 21-items questionnaire that ranges from a minimum of 0 points to a maximum of 63 points

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Don Carlo Gnocchi, Milan, MI, Italy